CLINICAL TRIAL: NCT05810129
Title: Effects of Crossed Education in Relation to Muscle Mass, Strength and Functionality in Patients Operated of Clavicular Fracture
Brief Title: Crossed Education in Relation to Muscle Mass in Patients Operated of Clavicular Fracture
Acronym: crossed1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de La Frontera (Other)
Responsible Party: Principal Investigator, Gabriel Nasri Marzuca-Nassr, PhD, Universidad de La Frontera
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 057/23
Record Dates: First submitted 2023-03-20; First posted 2023-04-12 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Clavicle Fracture
Keywords: muscle mass; cross education; eccentric training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: single-blind study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- standard physical therapy (Active Comparator): Men with clavicle fracture immobilized for 6 weeks + standard physical therapy for 12 weeks
  Interventions: Other: standard physical therapy
- concentric-eccentric strength training (Experimental): Men with clavicle fracture who perform concentric-eccentric strength training on the uninjured limb during the 6-week immobilization period + Posterior Standard PhysicalTherapy.
  Interventions: Other: concentric-eccentric strength training
- eccentric strength training (Experimental): Men with clavicle fracture who perform eccentric strength training on the unaffected limb during the 6-week period of immobilization + Posterior Standard Physical Therapy.
  Interventions: Other: eccentric strength training

INTERVENTIONS:
Other: concentric-eccentric strength training — Concentric-eccentric cross training in a 6-week immobilization period + 12-week standard kinesic therapy (2 times a week)
  Arms: concentric-eccentric strength training
Other: eccentric strength training — Eccentric cross training in immobilization period of 6 weeks + Standard kinesic therapy of 12 weeks (2 times a week)
  Arms: eccentric strength training
Other: standard physical therapy — Men with clavicle fracture immobilized for 6 weeks + standard physical therapy for 12 weeks
  Arms: standard physical therapy

SUMMARY:
The immobilization process after an operation or injury in the upper extremity causes a loss of muscle mass and strength of 0.2% and 1.3% per day, respectively. Currently, the use of cross-education, which is unilateral training in the uninjured limb, during the immobilization period, is expanding, demonstrating a magnitude of strength gain in the immobilized limb from 8% to 77% of the mean of strength of the trained limb. Despite the evidenced benefits of cross-education in unilateral injuries such as distal radius fracture, anterior cruciate ligament injury, and knee replacement, very little is known about this effect in shoulder immobilization after clavicle fracture.

DETAILED DESCRIPTION:
Objective: To determine the effectiveness of cross-education training through eccentric strength exercises compared to concentric-eccentric after the 6-week immobilization period and after 12 postoperative weeks in relation to muscle mass, strength, and functionality in patients operated of clavicular fracture.

Hypothesis: Cross-education training through eccentric strength exercises produces greater effects compared to concentric-eccentric training during the immobilization period and after 12 postoperative weeks, in relation to muscle mass, strength and functionality in patients operated for clavicle fracture.

Methodology: An experimental, randomized, single-blind study will be carried out, in which 39 men from 18 to 40 years of age will be recruited, who are awaiting surgery for clavicle fracture. They will be divided into three groups: control group (Standard Kinesic Therapy 12 weeks after immobilization of 6 weeks, n=13), concentric-eccentric group (concentric-eccentric strength training in the uninjured limb during the 6-week immobilization period + Standard Kinesics Therapy, n=13) and group eccentric (eccentric strength training on the uninjured limb during the 6-week immobilization period + Standard Kinesics Therapy, n=13).

Expected results: It is expected to observe a gain in muscle mass and strength in the trained limb and a maintenance/gain of muscle mass and strength in the groups that perform cross-training during the immobilization period, presenting the greatest benefit in the group that performs training eccentric force.

ELIGIBILITY:
Inclusion Criteria:

* Men from 18 to 40 years old, diagnosed with radiographically verified clavicle fracture and awaiting surgical procedure. They have a body mass index of not less than 18.5 and not more than 29.9 kg/m2 and sign an informed consent.

Exclusion Criteria:

* Patients with previous injuries, pathological fracture or polytrauma
* Patients who report pain, a history of rotator cuff tear or surgery in the non-injured upper extremity.
* Patients with uncontrolled cardiovascular diseases.
* Any history of neurological problems in the upper extremities.
* Use of nutritional supplementation (leucine, glutamine, casein, whey-protein, fatty acids and creatine) and/or Hormonal Replacement Therapy.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 39 (Estimated)
Dates: Start 2023-05-02 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Change in muscle thickness of the biceps brachii, triceps brachii and supraspinatus muscles by ultrasound. | before surgery, after 6 and 12 weeks postoperatively
  Change in muscle thickness of the biceps brachii, triceps brachii and supraspinatus muscles by ultrasound.

SECONDARY OUTCOMES:
Change in grip strength using a dynamometer and change in manual force at 90º elbow flexion, 45º shoulder flexion and 0º shoulder abduction | before surgery, after 6 and 12 weeks postoperatively
  Change in grip strength using a dynamometer and change in manual force at 90º elbow flexion, 45º shoulder flexion and 0º shoulder abduction
Upper and middle arm circumference change in both posterior arms | before surgery, after 6 and 12 weeks postoperatively
  Upper and middle arm circumference change in both posterior arms
Change in functionality using the Quick Dash questionnaire | before surgery, after 6 and 12 weeks postoperatively
  Change in functionality using the Quick Dash questionnaire
Change in relation to pain using the visual analogue scale | before surgery, after 6 and 12 weeks postoperatively
  Change in relation to pain using the visual analogue scale
Change in range of motion in elbow flexion, shoulder flexion, shoulder abduction, and rotations. | before surgery, after 6 and 12 weeks postoperatively
  Change in range of motion in elbow flexion, shoulder flexion, shoulder abduction, and rotations.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Marzuca, MSc, PhD, Principal Investigator — Universidad de La Frontera. Temuco, Chile
Locations (1):
- Universidad de La Frontera, Temuco, IX Región de La Araucanía, Chile